CLINICAL TRIAL: NCT06163027
Title: Effect of Shotblocker on Procedure-related Pain, Satisfaction and Comfort in Patients Receiving Spinal Anesthesia: Single-Blind, Randomized Controlled Study
Brief Title: Effect of Shotblocker on Procedure-related Pain, Satisfaction and Comfort in Patients Receiving Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tülay KILINÇ, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: tulay22
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Pain
Keywords: Spinal Anesthesia; Shotblocker; Pain; Satisfaction; Comfort
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shotblocker (Experimental): Shotblocker (experimental) group: Patients will undergo standard monitoring. The shotblocker will be sterilized before the procedure. Sterilization of the shotblocker will be controlled by the indicator on the packaging. Necessary sterilization conditions for spinal anesthesia application will be met and the procedure will be performed from the L3 -L4 or L4 -L5 spinal range. During the spinal anesthesia process, the protruding surface of the shot blocker will be placed in the area to be inserted, just before the spinal needle application. The shotblocker will be kept stationary throughout the procedure and pressure will continue to be applied. After entering for the spinal anesthesia procedure, the shot blocker will be removed. During the spinal anesthesia procedure, VAS, patient satisfaction and comfort scale will be applied to the patient in the first 1 minute and at the 24th hour after surgery.
  Interventions: Device: Shotblocker
- Placebo (Placebo Comparator): Placebo group: Patients will undergo standard monitoring (electrocardiogram, noninvasive blood pressure, peripheral oxygen saturation). The shotblocker will be sterilized before the procedure. Sterilization of the shotblocker will be controlled by the indicator on the packaging. Necessary sterilization conditions for spinal anesthesia application will be met and the procedure will be performed from the L3 -L4 or L4 -L5 spinal range. During the spinal anesthesia procedure, the reverse side of the shotblocker (without protrusions) will be placed on the skin surface and gently pressed with the fingertips. The shotblocker will be kept stationary throughout the procedure and pressure will continue to be applied. After entering for the spinal anesthesia procedure, the shot blocker will be removed. During the spinal anesthesia procedure, VAS, patient satisfaction and comfort scale will be applied to the patient in the first 1 minute and at the 24th hour after surgery.
  Interventions: Other: Shotblocker(Plasebo)
- Control (No Intervention): Routine treatment and care will be applied to the control group and no intervention will be made. During the spinal anesthesia procedure, VAS, patient satisfaction and comfort scale will be applied to the patient in the first 1 minute and at the 24th hour after surgery. The data obtained will be recorded in the patient diagnosis form. All interventions will be performed by the same anesthesiologist. The data will be filled in by a healthcare professional who is blinded to the study.

INTERVENTIONS:
Device: Shotblocker — Shotblocher will be administered during spinal needle injection
  Arms: Shotblocker
Other: Shotblocker(Plasebo) — The back side of the shotblocher will be applied during spinal needle injection
  Arms: Placebo

SUMMARY:
Although spinal anesthesia, which is increasingly common today, is a fast and reliable method, many patients are afraid of this procedure due to their fear of needles. Different methods have been studied to reduce pain during spinal needle insertion. One of the methods used to reduce pain due to needle insertion is ShotBlocker. This non-invasive, very simple to use application involves minimal risk and can be easily integrated into the application. For this reason, the research will be conducted to determine the effect of shot blockers on procedure-related pain, satisfaction and comfort in patients who will undergo spinal anesthesia.

DETAILED DESCRIPTION:
Spinal anesthesia is a type of anesthesia resulting from the injection of local anesthetic agents into the subarachnoid area and the blockade of the spinal nerve and dorsal root ganglia. It ensures that the patient is conscious during the operation, that spontaneous breathing continues, that the response to surgical stress is suppressed, that reflexes such as coughing and swallowing are preserved, that in addition to providing analgesia in the postoperative period, it provides rapid mobilization, facilitates the transition to early nutrition, is a low-cost technique, and has a short hospital stay. It is one of the most important advantages of spinal anesthesia. The rapid onset of effect and ease of application have made spinal anesthesia a widely preferred method in many interventions. However, most patients do not accept spinal anesthesia due to needle phobia.

The main reason for needle phobia, which is an important problem in anesthesia applications, is the occurrence of needle-related pain. Needle phobia and pain can also affect the quality of spinal anesthesia, making it difficult to administer and causing syncope.For this reason, methods such as EMLA cream, local anesthetic infiltration or application of EMLA cream before infiltration, local anesthesia application with a needle-free injection system, and vapocoolant spray are recommended to reduce superficial pain occurring under the skin / subcutaneous in spinal interventions. It has been reported that the application of local anesthetic infiltration before spinal anesthesia may cause pain during spinal needle insertion, sometimes not provide adequate analgesia, and may lead to the disappearance of anatomical signs. Local application of topical anesthetics such as EMLA cream is a painless method to reduce pain due to spinal needle insertion. However, it is recommended to apply it to the skin in a thick layer at least 30-90 minutes before the procedure to provide adequate analgesia. This situation causes various disadvantages regarding the use of EMLA cream to come to the fore. The requirement to apply it a certain time before the intervention limits its use in emergency cases. In elective cases, high and rapid patient circulation in the operating room makes it difficult to adjust the application time. Another disadvantage of EMLA cream is that it is costly. The use of local anesthetic infiltration with needle-free injection devices immediately before the procedure is also time-consuming and may interrupt the procedure and aseptic conditions if the lower or upper intervertebral space is needed for needle reinsertion. Therefore, a painless, effective and fast method is required. The shotblocker device is designed to reduce injection-related pain. ShotBlocker is reported to temporarily block peripheral nerve endings, preventing the perception and transmission of pain to the central nervous system, thus reducing pain. Pain, which is an undesirable experience for every patient, is defined as the fifth vital sign. Therefore, management of pain is very important regardless of whether it is acute or chronic. It is emphasized in the literature that the stress factors of anesthesia and surgery can be significantly reduced by relieving the pain that may occur due to various procedures. Additionally, patient satisfaction and comfort will increase. When the national and international literature was examined, only one study was found that used shotblockers to reduce pain due to spinal needle insertion. Therefore, the research was to be conducted to evaluate the effect of shot blockers on procedure-related pain, satisfaction and comfort in patients who will undergo spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Does not have a disease that may cause loss of sensation or loss of sensation
* Be open to communication
* Volunteering to participate in research

Exclusion Criteria:

* Experiencing a change in consciousness,
* Patients receiving centrally or peripherally acting analgesics or sedatives
* Patients with clinical conditions requiring urgent intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | up to 24 hours
  The visual analog scale will be used to assess the patient's pain intensity. It is a self-reported scale in the form of a 10- cm ruler indicating no pain at one end and unbearable pain at the other. Accordingly, the patient is told to evaluate his/ her pain between 0 and 10, with 0 indicating "no pain" and 10 indicating "unbearable pain

SECONDARY OUTCOMES:
Comfort Scale | up to 24 hours
  Comfort scale is a measuring tool that can be used horizontally and is 10 cm long. It starts with "most comfortable situation" and ends with "most uncomfortable situation". Patients are asked to rate their comfort level on a scale of 1 to 10.

OTHER OUTCOMES:
Visual Patient Satisfaction Scale | up to 24 hours
  The visual patient satisfaction scale consists of a 100 mm horizontal line without numbers on it. At one end of the line, "I am not satisfied at all"; At the other end, there is the phrase "I am very satisfied". With this scale, the patient is asked to determine his/her level of satisfaction with the care given and to mark the point on the line corresponding to his/her condition.